CLINICAL TRIAL: NCT02411604
Title: Expanded Access Study for Renal Transplant Patients With Envarsus XR™: Envarsus 3007
Brief Title: Expanded Access Study for Renal Transplant Patients With Envarsus XR ™
Status: Approved for marketing | Type: Expanded Access
Sponsor: Veloxis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: Envarsus® 3007
Record Dates: First submitted 2015-04-02; First posted 2015-04-08 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2015-12

CONDITIONS: Renal Failure
MeSH Terms: conditions — Renal Insufficiency | interventions — Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — Open label, multi-center, expanded access study for renal transplant patients with once daily Envarsus XR.
  Other Names: Envarsus XR

SUMMARY:
Open label, multi-center, expanded access study for renal transplant patients with once daily Envarsus XR (Tacrolimus).

DETAILED DESCRIPTION:
The study is designed to facilitate expanded access of Envarsus XR treatment to renal transplant patients. Patients are identified by the site investigator as a patient who has experienced favorable outcomes while in an Envarsus XR (LCP-Tacro) clinical study and/or the site investigator has identified a renal transplant patient with a medical need for an alternative tacrolimus treatment versus the patient's current tacrolimus treatment.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients will fulfill all of the following criteria:

  1. Patient age ≥18years old
  2. Willing to give written informed consent and is able to speak, write and understand English
  3. Patient understands potential risks or benefits with treatment of Envarsus XR
  4. Patients who have received a primary or secondary kidney transplant
  5. Patient who have received prior treatment with Envarsus XR (LCP-Tacro) and who are not currently participating in an Envarsus/LCP-Tacro study OR
  6. The treating Investigator has identified the patient as having a medical necessity for switching from their current tacrolimus treatment to Envarsus XR: Investigator is aware the medical necessity for switching is not related to the inability to purchase available tacrolimus.

Exclusion Criteria:

* Patients fulfilling any of the following criteria are NOT eligible for study inclusion:

  1. Recipients of organ transplants other than kidney
  2. Pregnant or nursing (lactating) women, or planning to become pregnant, where pregnancy is defined as a state of female after conception and until the termination of gestation, confirmed by a positive hCG serum or urine laboratory test.
  3. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant who are unwilling to use a defined SOC method of contraception, UNLESS they are
* Women whose career, lifestyle, or sexual orientation preclude intercourse with a male partner
* Women whose partners have been sterilized by vasectomy or other medically approved means

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult